CLINICAL TRIAL: NCT01139008
Title: Split-Face Tolerability Comparison Between MetroGel® (Metronidazole Gel) 1% Versus Finacea® (Azelaic Acid) Gel 15% in Subjects With Healthy Skin
Brief Title: Split-Face Tolerability Comparison Between MetroGel® 1% Versus Finacea® 15% in Subjects With Healthy Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10159
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2012-09

CONDITIONS: Skin Manifestations
MeSH Terms: conditions — Skin Manifestations | interventions — Metronidazole; Gels; azelaic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metronidazole 1% gel (Active Comparator)
  Interventions: Drug: metronidazole 1% gel
- azelaic acid 15% gel (Active Comparator)
  Interventions: Drug: azelaic acid 15% gel

INTERVENTIONS:
Drug: metronidazole 1% gel — Apply topically on one side of the face once daily for three weeks
  Other Names: MetroGel® 1%
  Arms: metronidazole 1% gel
Drug: azelaic acid 15% gel — Apply topically on the opposite side of the face twice daily for three weeks
  Other Names: Finacea® 15% Gel
  Arms: azelaic acid 15% gel

SUMMARY:
The purpose of this study is to compare the tolerability of MetroGel® (metronidazole gel) 1% to Finacea® (azelaic acid) Gel 15% in subjects with healthy skin applied according to product labeling for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults (ages 18 years or older)
* Subjects with healthy skin as determined by the clinical grader

Exclusion Criteria:

* Subjects with a degree of skin pigmentation that interferes with the reading of skin reactions
* Subjects with known allergy to one of the components of the study drugs (refer to the package inserts for MetroGel® 1% and Finacea® Gel 15%)
* Subjects who have participated in another investigational drug or device research study within 30 days of enrollment
* Subjects with a washout period for topical treatment on the treated area less than 1 week for corticosteroids and/or 4 weeks for retinoids
* Subjects with a washout period for systemic treatment less than 1 week for medications that may increase photosensitivity and/or 4 weeks for corticosteroids and/or 6 months for retinoids
* Subjects with current sunburn, eczema, atopic dermatitis, perioral dermatitis, rosacea, or other topical conditions on the area to be treated
* Subjects who foresee unprotected and intense UV exposure during the study (mountain sports, UV radiation, sunbathing, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Thomas J. Stephens and Associates, Inc., Carrollton, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on June 7, 2010 and the last subject was enrolled on June 7, 2010.
  Types of location: Investigative site was located at a research center.
Pre-assignment Details: Wash-out period up to baseline for topical treatment on the treated area was less than 1 week for corticosteroids and/or 4 weeks for retinoids; for systemic treatment less than 1 week for medications that may increase photosensitivity and/or 4 weeks for corticosteroids and/or 6 months for retinoids.
Groups:
- MetroGel® 1% and Finacea 15%: This was a randomized split-face study where metronidazole gel 1% was applied topically to one side of the face once daily for 3 weeks and azelaic acid gel 15% was applied to the opposite side of the face twice daily for 3 weeks
Period: Overall Study
Arm/Group | MetroGel® 1% and Finacea 15%
Started | 80
Completed | 74
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Non-compliant, lost product | 1

BASELINE CHARACTERISTICS:
Groups:
- MetroGel® 1% and Finacea® Gel 15%: This was a randomized split-face study where metronidazole gel 1% was applied topically to one side of the face once daily for 3 weeks and azelaic acid gel 15% was applied to the opposite side of the face twice daily for 3 weeks
Arm/Group | MetroGel® 1% and Finacea® Gel 15%
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were a Success With Regard to Worst Post-baseline Tolerability Assessment Scores in Each Assessment (Erythema, Scaling, Dryness, Stinging/Burning) From Baseline to Week 3
Description: Number of participants who were a success with regard to worst post-baseline tolerability assessment scores in each of the tolerability assessments at any time point between baseline and week 3. Tolerability assessments (erythema, scaling, dryness, stinging/burning) are evaluated on a scale from 0 - 4 (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) with 0 being best and 4 being worst. Success was defined as a tolerability score of 0.
Time Frame: baseline to week 3
Population: Safety
Measure: Number; unit: participants
Groups:
- MetroGel® 1%: metronidazole gel 1% - apply topically to one side of the face once daily for 3 weeks
- Finacea® Gel 15%: azelaic acid gel 15% - apply topically twice daily to the opposite side of the face
Arm/Group | MetroGel® 1% | Finacea® Gel 15%
Number analyzed (Participants) | 80 | 80
participants
  Erythema | 14 | 11
  Scaling | 79 | 78
  Dryness | 71 | 70
  Stinging/Burning | 72 | 65

2. Secondary Outcome: Number of Participants Who Were a Success With Regard to Worst-baseline Tolerability Assessment Scores in Each Assessment (Erythema, Scaling, Dryness, Stinging/Burning) on Day 22.
Description: Number of participants who were a success with regard to worst-baseline tolerability assessment scores for each assessment (erythema, scaling, dryness, stinging/burning) on day 22. Tolerability assessments (erythema, scaling, dryness, stinging/burning) are evaluated on a scale from 0 - 4 (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) with 0 being best and 4 being worst. Success was defined as a tolerability score of 0 for each assessment.
Time Frame: Day 22
Population: Safety
Measure: Number; unit: participants
Arm/Group | MetroGel® 1% | Finacea® Gel 15%
Number analyzed (Participants) | 80 | 80
participants
  Erythema | 34 | 29
  Scaling | 74 | 73
  Dryness | 73 | 73
  Stinging/Burning | 72 | 68

3. Secondary Outcome: 6 Question Subject Preference Survey at Week 3
Description: Number of participants per response to each question of the Subject Preference Survey at week 3
Time Frame: week 3
Population: Safety
Measure: Number; unit: participants
Groups:
- MetroGel® 1% and Finacea® Gel 15%: This is a split-face study where metronidazole gel 1% was applied topically to one side of the face once daily for 3 weeks and azelaic acid 15% gel was applied topically to the opposite side of the face twice daily for 3 weeks
Arm/Group | MetroGel® 1% and Finacea® Gel 15%
Number analyzed (Participants) | 80
participants
  1. Side of face felt better MetroGel® | 16
  1. Side of face felt better Finacea® | 20
  1. Side of face both felt same | 31
  1. Side of face neither felt better | 11
  1. Side of face Missing | 2
  2. Overall impression of MetroGel® Very pleasant | 16
  2. Overall impression of MetroGel® Pleasant | 25
  2. Overall impression of MetroGel® Okay | 32
  2. Overall impression of MetroGel® Unpleasant | 3
  2. Overall impression of MetroGel® Very Unpleasant | 2
  2. Overall impression of MetroGel® Missing | 2
  3. Overall impression of Finacea® Very pleasant | 15
  3. Overall impression of Finacea® Pleasant | 33
  3. Overall impression of Finacea® Okay | 25
  3. Overall impression of Finacea® Unpleasant | 4
  3. Overall impression of Finacea® Very unpleasant | 1
  3. Overall impression of Finacea® Missing | 2
  4. Side of face more sensitive MetroGel® | 12
  4. Side of face more sensitive Finacea® | 27
  4. Side of face more sensitive both felt same | 10
  4. Side of face more sensitive Neither | 29
  4. Side of face more sensitive Missing | 2
  5. Which side was easier to use MetroGel®? | 18
  5. Which side was easier to use Finacea®? | 21
  5. Which side was easier to use both equal? | 38
  5. Which side was easier to use Neither? | 1
  5. Which side was easier to use Missing | 2
  6. Which product tell a friend about MetroGel®? | 16
  6. Which product tell a friend about Finacea®? | 26
  6. Which product tell a friend about Both? | 25
  6. Which product tell a friend about Neither? | 11
  6. Which product tell a friend about Missing | 2

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), if applicable.
Arm/Group | MetroGel® 1% | Finacea® Gel 15%
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.